CLINICAL TRIAL: NCT05883280
Title: The Effect of Binaural Sound on the Occurrence of Emergence Delirium in Children Undergoing Strabismus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: pediatric ED_binaural beat
Record Dates: First submitted 2023-04-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binaural beats group (Experimental): Starting 30 minutes before the end of the surgery, a continuous pure tone binaural beat is delivered through headphones to the pediatric patient, with a frequency of 432 Hz in the left ear and 420 Hz in the right ear.
  Interventions: Other: Binaural beats
- Silence group (No Intervention): The headphones are placed on the pediatric patient, but there is no sound in the audio file being played.

INTERVENTIONS:
Other: Binaural beats — The binaural beat audio file consists of pure tones with a frequency of 432 Hz in the left ear and 420 Hz in the right ear. It is played through headphones starting 30 minutes before the end of the surgery.
  Arms: Binaural beats group

SUMMARY:
The hypothesis of this study is that providing continuous binaural beats with a phase difference in alpha frequency during anesthesia can reduce the incidence of emergence agitation in pediatric patients. To test this hypothesis, the occurrence of emergence agitation will be compared between the group that received binaural beats and the group that did not receive binaural beats.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 7 receiving a strabismus surgery under general anesthesia.
* American Society of Anesthesiologists Physical status classification 1-2.

Exclusion Criteria:

* Pediatric patients with hearing impairment or those who are currently using a hearing aid
* Pediatric patients with neurological disorders
* Pediatric patients with respiratory disorders

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence delirium in postanesthetic care unit (PACU) | within 1hr after the end of surgery

SECONDARY OUTCOMES:
Paediatric Assessment of Emergence Delirium (PAED) score | within 1hr after the end of surgery (every 10 minutes, the score will be checked)
Pain score (The Face, Legs, Activity, Cry and Consolability score) | within 1hr after the end of surgery
EEG analysis during emergence period | Time from discontinuation of sevoflurane to entering to PACU (within 1hr after the end of surgery)
  alpha, beta, gamma, delta, slow wave power and their ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park JB, Lee JH, Kim YJ, Lee DJ, Seo JH. The Effect of Binaural Sound on the Occurrence of Emergence Delirium in Children Undergoing Strabismus Surgery: A Randomized Controlled Trial. Paediatr Anaesth. 2026 Feb 6. doi: 10.1002/pan.70137. Online ahead of print. PMID 41646000